CLINICAL TRIAL: NCT04457856
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Single Ascending Dose and Multiple Ascending Doses of TJ003234 in Rheumatoid Arthritis Patients
Brief Title: A Study of TJ003234 in Rheumatoid Arthritis Patients
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: I-Mab Biopharma US Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TJ003234RAR102
Record Dates: First submitted 2020-06-28; First posted 2020-07-07 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; biologics
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — plonmarlimab

STUDY DESIGN:
Intervention Model Description: Randomized, Double-blind, Placebo-controlled
Who Masked: Participant
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TJ003234 (Experimental): Intravenous administration, single dose (0.3-1-3-10mg/kg) or multiple dose (1-3-6mg/kg, once every week, for 8 weeks) Mode of administration: The investigational drug is administered by intravenous infusion
  Interventions: Biological: TJ003234 injection
- Placebo (Placebo Comparator): Intravenous administration, single dose (0.3-1-3-10mg/kg) or multiple dose (1-3-6mg/kg, once every week, for 8 weeks) Mode of administration: The investigational drug is administered by intravenous infusion
  Interventions: Biological: TJ003234 injection

INTERVENTIONS:
Biological: TJ003234 injection — Intravenous administration, single dose (0.3-1-3-10mg/kg) or multiple dose (1-3-6mg/kg, once every week, for 8 weeks)

SUMMARY:
Study Purpose and Design: A Multi-center, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Single Ascending Dose and Multiple Ascending Doses of TJ003234 in Rheumatoid Arthritis Patients.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be ≥ 18 and ≤70 years old when signing the informed consent, with no limitation of gender.
* Established Rheumatoid arthritis patients, diagnosed by ACR/EULAR criteria 2010 at least 6 months prior to randomisation.
* Single Ascending Dose: DAS28 score≤3.2. Multiple Ascending Dose: DAS28 score≤5.1 and >3.2.
* Allowed one or more standard treatments, but the start date should no later than 12 weeks(84 days) before the randomisation and should take at a stable dose more than 4 weeks(28 days) before the randomisation. The combination taken of Methotrexate (MTX) and leflunomide was not allowed within 4 weeks (28 days) before randomization.
* Subjects must agree to attendance the study and signed the inform concent by themselves.
* Subjects(include subjects's wife) are no pregnancy plan during the sceering and 3 months after complete the study and agree to use contraceptives that protocol suggest.

Exclusion Criteria:

* Employees of the hospital or any other person that paticipant in the study and their immedidte family members.
* A documented history of an autoimmune disease other than RA (other than secondary Sjögren's syndrome) .
* Previous received Any biologic DMARD therapy including tsDMARD. •A positive hepatitis B (HBsAg, anti-HBc, and/or IgM anti-HBc), hepatitis C or HIV test at screening, indicative of a current or past infection.
* A history of active tuberculosis (TB) or positive serological test for TB (Quantiferon TB Gold or T-SPOT).
* Female patients who are pregnant during the study, or are breastfeeding. •Malignancy, or prior malignancy, with a disease free interval of <5 years after diagnosis and intervention except curative treatment for basal and squamous cell skin cancer.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2020-08-06 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Number of subject with adverse events(AEs) | First dose up to last follow-up visit (i.e. 90 days after dosing for single dose part, 140 days after first dose for multiple dose part)
  Number of subject with adverse events(AEs) to evaluate satety in patient with RA with vital signs, Electrocardiograms, physical examinations, laboratory tests and respiratory-related examinations

SECONDARY OUTCOMES:
AUC from time 0 to the time of the last quantifiable concentration AUC0-tlast of TJ003234 | Day1 to 90 days after dosing for single dose part, 140 days after for multiple dose part
  AUC from time 0 to the time of the last quantifiable concentration AUC0-tlast of TJ003234
Maximum observed plasma concentration (Cmax) of TJ003234 | Day1 to 90 days after dosing for single dose part, 140 days after for multiple dose part
  Maximum observed plasma concentration (Cmax) of TJ003234
The proportion of subjects who produce anti-drug antibodies | Day1 to 90 days after dosing for single dose part, 140 days after for multiple dose part
  The proportion of subjects who produce anti-drug antibodies
The proportion of subjects who produce neutralizing antibodies | Day1 to 90 days after dosing for single dose part, 140 days after for multiple dose part
  The proportion of subjects who produce neutralizing antibodies
The proportion of subjects who produce the titers of anti-drug antibodies and neutralizing antibodies | Day1 to 90 days after dosing for single dose part, 140 days after for multiple dose part
  The proportion of subjects who produce the titers of anti-drug antibodies and neutralizing antibodies

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - The first affiliated hospital of bengbu medical college, Bengbu, Anhui
  - Peking university people's Hospital, Beijing, Beijing Municipality
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - Zhongda Hospital southeast university, Nanjing, Jiangsu
  - FuDan University shanghai huashan Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No